CLINICAL TRIAL: NCT01151956
Title: Actinic Keratoses and 5% Topical Imiquimod: Lessons to Learn From a Prospective Non-Interventional Study by 93 Office-based Dermatologists
Brief Title: Imiquimod and Actinic Keratoses: an Observational Study
Status: Completed | Type: Observational
Sponsor: Federal University Teaching Hospital, Feldkirch, Austria (Other)
Collaborators: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Dr. Lydia Schuster, Meda Pharma Austria
Other Study IDs: OBIMQ465-AK-08
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2008-04

CONDITIONS: Actinic Keratosis
Keywords: observational study; actinic keratosis; imiquimod
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- actinic keratosis patients: patients who see their non-hospital based dermatologist, because of multiple actinic keratoses and who are then routinely treated with topical 5% Imiquimod

SUMMARY:
Objective: To show how dermatologists treat actinic keratoses with imiquimod 5% cream in their daily clinical routine.

Design: Prospective, non-interventional, observational, multicenter clinical study.

Setting: Offices of 93 non hospital based Austrian dermatologists. Participants: Inclusion of the 463 patients into the study was solely based on the treatment decision of the dermatologist and the patients will.

Interventions: No specific interventions except suggested time points of visits with pre-defined documentation forms. The therapy of actinic keratoses followed the imiquimod label (3x/week for 4 weeks, 4 therapy free weeks, another 3x/week for 4 weeks, when needed) Main outcome measure: Information about the typical imiquimod patient, therapeutic course, treatment decisions, safety and satisfaction of patients/dermatologists.

DETAILED DESCRIPTION:
DESIGN AND STUDY POPULATION The present study was a prospective, open label, non interventional clinical study precisely documenting the routine therapy of AK with imiquimod 5% cream. According to Austrian regulations, for an observational study where medication follows the label of the drug it is not necessary to seek approval from the federal ethic committee. Except the presence of multiple AK there were no further rules to include the patient into the study. Following the dermatologists decision and the patients will, 463 patients were treated in the offices of 93 non hospital based Austrian dermatologists. There were no further interventions except recommended time points of visits documented with pre-defined forms. Imiquimod therapy followed the label. Patients applied imiquimod at home 3x/week (typically Monday, Wednesday and Thursday) for 4 weeks, followed by 4 therapy free weeks and another 3x/week 4 weeks therapeutic course, when needed. Recommended visits (V) were: V1 baseline, week 0; V2, week 4 (end of the first treatment cycle); V3, week 8 (decision point for the need of a second treatment course); V4, week 16 (for those receiving a second treatment course). Additional unplanned visits (VX) were possible and also documented.

STUDY PROCEDURES At baseline patients characteristics, i.e. sex, age, size and weight were documented together with the information who referred the patient to the dermatologist. Next, the patient skin cancer family history and the AK history including the time of the first presentation as well as former therapies and their success were asked. This was followed by a dermatological examination which defined the numbers of AK lesions, their location and the nature as well as intensity of initial skin signs (erosion, crusting, erythema, ulceration, swelling, others, graded as no, mild, moderate, severe). Before the start of the therapy, patients were informed about the typical imiquimod skin reactions by a set of pictures and a brochure. In addition, all patients got a treatment plan showing the different phases of the therapy and the time points when imiquimod should be applied. Within this plan patients also had the possibility to document their imiquimod use. Also at baseline, potential systemic and local co-medications were documented.

At all following visits, nature and intensity of Imiquimod related skin responses potential adverse events and pre-final termination of the study were acknowledged. Decisions by the dermatologists were documented as (i) nature of the topical post imiquimod treatment of therapeutic skin reactions (V2, V3, V4, VX), (ii) initiation of a second therapeutic course, or character of the alternative therapy (V3) as well as (iii) full clearing of all lesions, or number of remaining lesions (V3, V4). At VX the dermatologist reaction to this unplanned visit was asked (no consequences, temporary discontinuation of the therapy - how long, topical treatment of the therapy related skin symptoms, or, pre-final termination of the therapy). At the end of the study, reasons for a potential pre-final termination (lack of efficacy, patients wish, adverse events, others), the kind of subsequent therapy for remaining AK lesions, satisfaction of the dermatologist with the efficacy, tolerability and the cosmetic outcome of the imiquimod therapy as well as patients general and specific satisfaction with the cosmetic outcome and his estimation about the therapy success including his grade of relief with the solved problem were delineated.

ELIGIBILITY:
Inclusion Criteria:

* no study specific, just following the label of imiquimod

Exclusion Criteria:

* no study specific, just following the label of Imiquimod

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with actinic keratoses who are routinely treated with topical 5% Imiquimod by non-hospital based dermatologists
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2008-05; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Management of the actic keratosis patient routinely treated with Imiquimod by non-hospital based dermatologists | 12 weeks
  Information about the typical imiquimod patient, therapeutic course, treatment decisions and satisfaction of patients/dermatologists.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Strohal, AssocProfDr, Principal Investigator — Federal University Teaching Hospital of Feldkirch, Dept. of Dermatology

REFERENCES:
- [Derived] Strohal R, Kerl H, Schuster L. Treatment of actinic keratoses with 5% topical imiquimod: a multicenter prospective observational study from 93 Austrian office-based dermatologists. J Drugs Dermatol. 2012 May;11(5):574-8. PMID 22527424